CLINICAL TRIAL: NCT05510063
Title: A Phase IV, Randomized, Double-blind, Parallel-group, Multiple-dose, Active Comparator, Multicenter Clinical Study to Evaluate the Pharmacokinetics, Efficacy, Safety, and Immunogenicity of SB5 Versus Humira in Subjects With Moderate to Severe Chronic Plaque Psoriasis
Brief Title: Pharmacokinetics, Efficacy, Safety, and Immunogenicity of SB5 Versus Humira in Subjects With Moderate to Severe Chronic Plaque Psoriasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Samsung Bioepis Co., Ltd. (Industry)
Collaborators: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SB5-4001
Record Dates: First submitted 2022-08-19; First posted 2022-08-22 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Plaque Psoriasis
Keywords: Psoriasis; Adalimumab
MeSH Terms: conditions — Psoriasis | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Switched between Humira and SB5 (Experimental): All subjects will receive an initial dose of Humira 80 mg at Week 0, followed by Humira 40 mg every other week starting one week after the initial dose up to Week 11. From Week 13, the subjects will switch between Humira and SB5 up to Week 23.
  Interventions: Drug: Humira (Adalimumab); Drug: SB5 (Adalimumab Biosimilar)
- Continued on Humira (Active Comparator): All subjects will receive an initial dose of Humira 80 mg at Week 0, followed by Humira 40 mg every other week starting one week after the initial dose up to Week 23.
  Interventions: Drug: Humira (Adalimumab)

INTERVENTIONS:
Drug: Humira (Adalimumab) — Subcutaneous (SC) injection
Drug: SB5 (Adalimumab Biosimilar) — Subcutaneous (SC) injection
  Arms: Switched between Humira and SB5

SUMMARY:
This is a Phase IV, randomized, double-blind, parallel-group, multiple-dose, active comparator, multicenter clinical study to evaluate the pharmacokinetics, efficacy, safety, and immunogenicity of SB5 versus Humira in subjects with moderate to severe chronic plaque psoriasis.

DETAILED DESCRIPTION:
The primary objective of this study is to assess the pharmacokinetic similarity in subjects with moderate to severe plaque psoriasis who switch between Humira and SB5 to those receiving Humira continuously.

All entered subjects will be treated with Humira during a lead-in period of 13 weeks. At Week 13, subjects who achieved at least a 50% reduction in Psoriasis Area and Severity Index (PASI50) response will be randomized in a 1:1 ratio to either be switched between Humira and SB5 or continue on Humira.

ELIGIBILITY:
Inclusion Criteria:

* Have no history of Adalimumab and cell-depleting biologics
* Have no history of any other biologics use within 6 months prior to Week 0
* Have plaque psoriasis diagnosed at least 6 months, with or without psoriatic arthritis
* Have plaque psoriasis with the involvement and severity of total affected BSA ≥ 10%, PASI score of ≥ 12 and PGA score of ≥ 3 (moderate)
* Considered to be a candidate for phototherapy or systemic therapy for psoriasis
* Adequate hematological, renal, and hepatic function by central lab
* Non-childbearing potential female, or childbearing potential female subjects or male subjects with their partners who agree to use at least two forms of appropriate contraception method from Screening until 5 months after the last dose of IP

Exclusion Criteria:

* Have nonplaque forms of psoriasis, including erythrodermic, pustular, guttate, or drug-induced psoriasis
* Have other skin disease than psoriasis that requires topical, phototherapy or systemic therapy
* Known allergic reactions or hypersensitivity to adalimumab or to any ingredients of SB5 or Humira
* Have received phototherapy or conventional systemic therapy within 4 weeks prior to Week 0
* Have received topical therapy for psoriasis within 2 weeks prior to Week 0, however class 6/7 corticosteroids are allowed on face and groin
* Women who are pregnant or nursing at Screening, or men and women planning pregnancy during the study period and until 5 months after the last dose of IP
* Have received a live or live attenuated viral vaccine or a live bacterial vaccine within 8 weeks prior to Week 0. Non-live COVID-19 vaccines are allowed
* Have active or latent tuberculosis
* History of ongoing infection or a positive test of HBV, HCV, or HIV infection
* History of sepsis, chronic or recurrent infection
* History of lymphoproliferative disease or leukaemia
* History of malignancy within the last 5 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 371 (Actual)
Dates: Start 2022-08-04 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-05-04 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve over the dosing interval (AUCtau) | Week 23 to Week 25
Maximum serum concentration during the dosing interval (Cmax) | Week 23 to Week 25

CONTACTS AND LOCATIONS:
Locations (23):
- Bulgaria (3):
  - SB Investigative Site, Dupnitsa
  - SB Investigative Site, Pleven
  - SB Investigative Site, Sofia
- Czechia (3):
  - SB Investigative Site, Ostrava
  - SB Investigative Site, Pardubice
  - SB Investigative Site, Prague
- Lithuania (2):
  - SB Investigative Site, Kaunas
  - SB Investigative Site, Vilnius
- Poland (15):
  - SB Investigative Site, Bialystok
  - SB Investigative Site, Bydgoszcz
  - SB Investigative Site, Gdansk
  - SB Investigative Site, Gdynia
  - SB Investigative Site, Krakow
  - SB Investigative Site, Lodz
  - SB Investigative Site, Lublin
  - SB Investigative Site, Nowa Sól
  - SB Investigative Site, Olsztyn
  - SB Investigative Site, Osielsko
  - SB Investigative Site, Poznan
  - SB Investigative Site, Siedlce
  - SB Investigative Site, Szczecin
  - SB Investigative Site, Świdnik
  - SB Investigative Site, Warsaw